CLINICAL TRIAL: NCT01844596
Title: Optimizing Linkage and Retention to Hypertension Care in Rural Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 11-1056
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Hypertension; High Blood Pressure
Keywords: linkage to care; hypertension management; behavioral science; cardiovascular health; global health; multi-disciplinary implementation research approach; linking and retaining; community health workers; CHWs; behavioral communication strategy; smartphone-based tool; electronic health record; retention to care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Usual Care: Community Health Workers (CHW) with standard training on recruitment of individuals.
- behavioral communication strategy (Experimental): Community Health Workers with an additional tailored behavioral communication strategy.
  Interventions: Behavioral: behavioral communication strategy
- Behavioral communication strategy, plus smartphone-based tool (Experimental): Community Health Workers with a tailored behavioral communication strategy, also equipped with smartphone-based tool linked to the AMPATH Medical Record System (AMRS).
  Interventions: Behavioral: Behavioral communication strategy, plus smartphone-based tool

INTERVENTIONS:
Behavioral: behavioral communication strategy — Community Health Workers with an additional tailored behavioral communication strategy.
  Arms: behavioral communication strategy
Behavioral: Behavioral communication strategy, plus smartphone-based tool — Community Health Workers with a tailored behavioral communication strategy, also equipped with smartphone-based tool linked to the AMPATH Medical Record System (AMRS).
  Arms: Behavioral communication strategy, plus smartphone-based tool

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in sub-Saharan Africa among adults above age 30. The prevalence of hypertension, a major risk factor for CVD, is increasing over time in sub-Saharan Africa, exerting a significant epidemiologic and economic burden on the region. Without adequate control of hypertension, its health and economic burden will increase drastically in the decades ahead. Well established and evidence-based interventions to manage hypertension exist; however, treatment and control rates are low.

A critical component of hypertension management is to facilitate sustained access of affected individuals to effective clinical services. In partnership with the Government of Kenya, the United States Agency for International Development-Academic Model Providing Access to Healthcare Partnership (AMPATH) is expanding its clinical scope of work in rural western Kenya to include hypertension and other chronic diseases.

However, linking and retaining individuals with elevated blood pressure to the clinical care program has been difficult. Thus, the overall objective of this application is to utilize a multi-disciplinary implementation research approach to address the challenge of linking and retaining hypertensive individuals to a hypertension management program. We aim to add to existing knowledge on scalable and sustainable strategies for optimizing control of hypertension and other chronic diseases in low- and middle-income countries.

DETAILED DESCRIPTION:
Hypertension awareness, treatment, and control rates are low in most regions of the world. A critical component of hypertension management is to facilitate sustained access of affected individuals to effective clinical services. In partnership with the Government of Kenya, the Academic Model Providing Access to Healthcare (AMPATH) Partnership is expanding its clinical scope of work in rural western Kenya to include hypertension and other chronic diseases. However, linking and retaining individuals with elevated blood pressure to the clinical care program has been difficult. To address this challenge, we propose to develop and evaluate innovative community-based strategies and initiatives supported by mobile technology.

The objective of this application is to utilize a multi-disciplinary implementation research approach to address the challenge of linking and retaining hypertensive individuals to a hypertension management program. The central hypothesis is: community health workers (CHWs), equipped with a tailored behavioral communication strategy and a smartphone-based tool linked to an electronic health record, can increase linkage and retention of hypertensive individuals to a hypertension care program and thereby significantly reduce blood pressure among these patients. We further hypothesize that these interventions will be cost-effective.

This research will generate innovative and productive solutions to the expanding global problem of hypertension, and will add to existing knowledge on scalable and sustainable strategies for effectively managing hypertension and other chronic diseases in low- and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* elevated BP (SBP > 140 or DBP >90)

Exclusion Criteria:

* acutely ill and require immediate medical attention at the time of home-based testing
* individuals who do not provide informed consent during home-based testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1455 (Actual)
Dates: Start 2014-04; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Documented linkage to care following home-based testing | up to 5 years
  An individual who links to care on his/her own within one month of home-based blood pressure testing will be characterized as "self-linked" or after a community health worker (CHW) visit, sh/he will be characterized as "CHW-mediated linked."
One year change in systolic blood pressure among hypertensive individuals | up to one year
  One year change in systolic blood pressure among hypertensive individuals.

SECONDARY OUTCOMES:
Blood Pressure controlled | up to 5 years
  Percentage of hypertensive individuals whose BP is controlled (<140/90) at the final clinic visit
Medication adherence | up to 5 years
  Medication adherence will be defined as number of doses taken divided by number of doses prescribed, for the previous one month.
behavioral changes | up to 5 years
  Behavioral changes include physical activity, diet (salt, fruit/vegetable intake), and tobacco use.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Moi University School of Medicine, Eldoret, Kenya

REFERENCES:
- [Derived] Vedanthan R, Kamano JH, DeLong AK, Naanyu V, Binanay CA, Bloomfield GS, Chrysanthopoulou SA, Finkelstein EA, Hogan JW, Horowitz CR, Inui TS, Menya D, Orango V, Velazquez EJ, Were MC, Kimaiyo S, Fuster V. Community Health Workers Improve Linkage to Hypertension Care in Western Kenya. J Am Coll Cardiol. 2019 Oct 15;74(15):1897-1906. doi: 10.1016/j.jacc.2019.08.003. Epub 2019 Sep 2. PMID 31487546
- [Derived] Vedanthan R, Kamano JH, Naanyu V, Delong AK, Were MC, Finkelstein EA, Menya D, Akwanalo CO, Bloomfield GS, Binanay CA, Velazquez EJ, Hogan JW, Horowitz CR, Inui TS, Kimaiyo S, Fuster V. Optimizing linkage and retention to hypertension care in rural Kenya (LARK hypertension study): study protocol for a randomized controlled trial. Trials. 2014 Apr 27;15:143. doi: 10.1186/1745-6215-15-143. PMID 24767476